CLINICAL TRIAL: NCT00079742
Title: A Phase II, Multicenter, Randomized, Controlled, Open-Label Study of the Safety and Efficacy of Nutropin AQ [Somatropin (DNA Origin) Injection] for the Treatment of Growth Restriction in Children With Cystic Fibrosis
Brief Title: A Study to Evaluate Nutropin AQ for the Treatment of Growth Restriction in Children With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Purpose: Treatment
Other Study IDs: L2762g
Record Dates: First submitted 2004-03-11; First posted 2004-03-16 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Cystic Fibrosis
Keywords: Growth restriction in children with cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Growth Hormone; Human Growth Hormone; Injections

INTERVENTIONS:
Drug: Nutropin AQ [somatropin (DNA origin) injection]

SUMMARY:
This is a Phase II, multicenter, randomized, controlled, open-label trial of the safety and efficacy of Nutropin AQ administered subcutaneously (SC) daily in prepubertal children with CF and growth restriction.

ELIGIBILITY:
Inclusion Criteria:

* Ability of parent or legal guardian to provide written informed consent and, if applicable, pediatric assent and compliance with study assessments for the full duration of the study
* Diagnosis of CF by sweat or genetic testing
* Between the ages of 5 and 12 years for girls and 5 and 13 years for boys
* Ability to perform pulmonary function tests in a reproducible manner, per American Thoracic Society guidelines for spirometry
* Height <= 10th percentile for age and sex
* Prepubertal, Tanner Stage 1
* Bone age of the non-dominant hand and wrist obtained no more than 6 months prior to study entry (bone age must be <= 10 years for girls and <= 11 years for boys as read using the method of Greulich and Pyle)
* Adequate caloric intake (following the CFF guidelines is encouraged; caloric intake must be documented at screening using a 24-hour food diary)
* Normal thyroid function

Exclusion Criteria:

* Prior or current rhGH use
* History of short stature due to GHD
* History within the 12 months prior to screening of glucose intolerance (impaired glucose tolerance) or CF-related diabetes (CFRD) as defined by at least one of the following: fasting serum glucose of >= 126 mg/dL on two or more occasions; fasting serum glucose of >= 126 mg/dL plus any casual (previously called random) glucose level >= 200 mg/dL; casual (previously called random) glucose of >= 200 mg/dL on two or more occasions; fasting serum glucose of <= 126 mg/dL but 2-hour post oral glucose load of 140-199 mg/dL (impaired glucose tolerance) on two or more occasions; if a subject meets the criteria for impaired glucose tolerance or CFRD in the screening glucose tolerance test, even if there is no history of impaired glucose tolerance, the subject will not be eligible for the study.
* Infection with Burkholderia cepacia
* Qualitative change in antibiotic treatment (e.g., for exacerbation of lung infection) within 14 days of study entry
* Hospitalization or treatment with systemic corticosteroids during the 30 days prior to study entry
* Inability to adhere to previously documented adequate nutrition
* Active neoplasia
* Participation in any other investigational study (including investigational drug studies) within 30 days of enrollment or during the study if in the treatment arm, except for participation in observational and questionnaire studies (untreated)
* Subjects who require, as part of the their medical care, scheduled elective hospitalizations for IV antibiotic therapy

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2003-09; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To determine the safety and efficacy of Nutropin AQ in treating growth restriction and increasing lean body mass (LBM) in children with cystic fibrosis (CF) and growth restriction.

SECONDARY OUTCOMES:
To evaluate the effects of Nutropin AQ treatment on pulmonary function, disease-related exacerbations, and exercise tolerance in children with CF and growth restriction.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lippe, M.D., Study Director — Genentech, Inc.